CLINICAL TRIAL: NCT06872216
Title: Evaluation the Impact of Dry Cupping Therapy on Microvascular Reactivity by Near-infrared Spectroscopy with Vascular Occlusion Test in Healthy Volunteers
Brief Title: Effect of Cupping Therapy on Microcirculation in Healthy Volunteers
Acronym: CTWN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NIRS-CUPPİNG
Record Dates: First submitted 2025-02-18; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Microcirculation
Keywords: Cupping therapy; microcirculation; near-infrared spectroscopy
MeSH Terms: interventions — Cupping Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cupping therapy (Other): nırs monitored during vot test pre-post cupping therapy
  Interventions: Procedure: cupping therapy; Diagnostic Test: Vascular occlusion test

INTERVENTIONS:
Procedure: cupping therapy — After the initial vascular occlusion test and a subsequent 10-minute rest period, the plastic therapy cup was placed on the forearm, 5 cm away from the medial and lateral epicondyles by a certified cupping therapist. The size of used cup was determined according to the size of the volunteer's forearm which cover 50% of the area. The cup was vacuumed two times full pumping with a manual hand pump and remained in place for 5 minutes. And then the air was removed by releasing the cups through the release valve.
Diagnostic Test: Vascular occlusion test — A blood pressure cuff was placed on the upper arm. The adult probe of the NIRS device (Covidien INVOS™ 5100C Cerebral/Somatic Oximeter, Dublin) was placed on the thenar region of the ipsilateral hand and the regional oxygen value was recorded during all study term. Baseline arterial pressure and oxygen saturation were monitored (GE Healthcare Oy, Helsinki, Finland) from the side of dominant hand and recorded. After a 3-minute stabilization period, the vascular occlusion protocol was started. The blood pressure cuff was rapidly inflated within 3-4 seconds to 50 mmHg above baseline systolic blood pressure and kept at this pressure during 3 minutes. Following this, the cuff was deflated within 1 second. Five minutes after cupping therapy this protocol had done again.

SUMMARY:
Twenty healthy volunteers were included in the study. The NIRS was placed on the thenar region of the hand. The vascular occlusion protocol had been done before and after cupping therapy (CT). Regional oxygen saturation (rSO2), the times to the lowest and highest values were recorded. The occlusion slope, the recovery slope and the first 10 second recovery slope were calculated.

DETAILED DESCRIPTION:
Participants rested in a seated position at standard temperature for at least 10 minutes. A blood pressure cuff was applied to the upper arm, and the NIRS device (Covidien INVOS™ 5100C Cerebral/Somatic Oximeter, Dublin) was used to monitor regional oxygen levels in the thenar region of the hand throughout the protocol. After a 3-minute stabilization period, the vascular occlusion protocol commenced: the blood pressure cuff was inflated rapidly within 3-4 seconds to 50 mmHg above the baseline systolic blood pressure and maintained for 3 minutes, then deflated within 1 second. The participant rested for another 10 minutes before a certified cupping therapist placed a plastic therapy cup on the forearm, 5 cm from the medial and lateral epicondyles. The size of the cup was based on the participant's forearm, covering 50% of the area. The cup was vacuumed twice using a manual hand pump and left in place for 5 minutes before the air was released through the valve. Following a 3-minute stabilization period, the vascular occlusion protocol was repeated. During the test, rSO2 values and the time to reach the lowest and highest values were recorded. Using this data, the occlusion slope, recovery slope, and 10-second recovery slope were calculated. The occlusion slope was determined by the formula [(baseline rSO2 - minimum rSO2) / time to lowest rSO2], in %/minute. The recovery slope was calculated as [(minimum rSO2 - maximum rSO2) / time to reach the highest rSO2], in %/second. The 10-second recovery slope was calculated as [(minimum rSO2 - rSO2 at 10 seconds) / 10 seconds].

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Healthy

Exclusion Criteria:

* Smoking or using tobacco products
* Taking alcohol or other substances, or any medication
* Have conditions affecting microcirculation
* Have acute or chronic pain
* Anemia
* Obesity
* Reynaud's phenomenon
* Baseline blood pressure being 140-90mmHg or above
* sPO2 value being below 96%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
the rSO2 values | Periprocedural
  monitored at tenar region on the dominant hand with near infrared spectrometry

SECONDARY OUTCOMES:
the time to reach the lowest rSO2 | Periprocedural
  the interval of the basal and minimal rSO2 is measured
the time to reach the highest values | Periprocedural
  the interval of the minimal to maximal rSO2 is measured
the occlusion slope | Periprocedural
  The occlusion slope was calculated based on time to reach to the lowest rSO2 as [(baseline rSO2 -minimum rSO2)/ time to lowest rSO2], %/minute.
Recovery slope | Periprocedural
  Recovery slope was calculated based on the time to reach the highest rSO2 value as [(minimum rSO2 - maximum rSO2)/ time to reach the highest rSO2], %/second.
The 10th second recovery slope | Periprocedural
  The 10th second recovery slope was calculated as [(minimum rSO2 - at first 10th second rSO2)/ 10 second].

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa üniversity, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu W, Piao S, Meng Xi, Wei L. Effects of cupping on blood flow under skin of back in healthy human. World Journal of Acupuncture - Moxibustion. 2013; 23 (3): 50-52. doi.org/10.1016/S1003-5257(13)60061-6.
- [Background] Gomez H, Torres A, Polanco P, Kim HK, Zenker S, Puyana JC, Pinsky MR. Use of non-invasive NIRS during a vascular occlusion test to assess dynamic tissue O(2) saturation response. Intensive Care Med. 2008 Sep;34(9):1600-7. doi: 10.1007/s00134-008-1145-1. Epub 2008 Jun 4. PMID 18523754